CLINICAL TRIAL: NCT04298424
Title: Effects of the Peer-Led Self-Management Program (PLSM) on Self-Efficacy, Self-Management and Physiological Measures Among Elderly Patients With Diabetes: Pilot Randomized Controlled Trial
Brief Title: the Peer-Led Self-Management Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 17B-023
Record Dates: First submitted 2020-02-18; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Self-Efficacy; Self-Management; Older Adults; Diabetes
Keywords: Diabetes Mellitus; Older; Self-Efficacy, Self-Management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-led (Experimental): The experimental group will conduct a 4-week peer self-management program and receive the original outpatient routine care.
  Interventions: Other: PLSM
- No Peer-led (No Intervention): The control group will only issue a self-management manual and receive the original outpatient routine care.

INTERVENTIONS:
Other: PLSM — The program was designed for implementation over 4 consecutive weeks, with groups of 6-8 people each attending one 60-90-minute class per week. Peer leaders lead the groups to promote interaction, sharing, and support, and assist in goal setting to address behavior-related health problems, and thereby the development and implementation of strategies to achieve suitable, sustainable, and feasible self-management behavior.
  Arms: Peer-led

SUMMARY:
Elderly patients have the deficiency of motivation and confidence in self-management that are mainly influenced by physiological function, social psychology, emotion and low health literacy, resulting in poor self-management and glycemic control. According to the study, elderly patients can learn the skill of self-management more effectively through the peer leaders who have the same culture background, the life experience in disease care and the successful self-management experiences. The Self-Management Program of diabetes for the elderly will be in progress with the peer leadership concept.( the Peer-Led Self-Management Program). The aim of the pilot study was to explore the feasibility and effects of the Peer-Led Self-Management Program (PLSM).

This pilot study uses two groups of block randomized controlled trials with pretest and posttest study. The test group will conduct a four-week Peer-Led Self-Management Program and the general outpatient care while the control group will implement the general outpatient care. In this study, the physiological parameters of Diabetes were used to evaluate the difference between the pre-and post-intervention measures.

DETAILED DESCRIPTION:
Most current self-management programs are developed for implementation by healthcare professionals. These professionals cannot fully perceive disease management needs and obstacles of older adults due to a lack of similar illness experience. To develop a self-management training program for older adult peer leaders with diabetes and to assess its feasibility.

This study was conducted in three stages. In stage 1, the peer leader training program was developed using experiential learning theory as the framework and self-regulation theory as the strategy for activity design. The 4-week training program was implemented for 4 hours/week. In stage 2, the feasibility of the training program was assessed. A peer leader training assessment tool was developed and used to evaluate peer leaders' leadership skills for self-management programs. Peer leaders' attendance rate and their viewpoints toward the training program through qualitative interview, willingness to lead self-management programs for older adults with diabetes in the community in the future were also assessed. In stage 3, This pilot study will take elderly diabetic patients in a community health station in Taiwan. The program will be conducted by peer leaders who have completed training to lead elderly diabetic patients and promote interaction, sharing, and support among peers. Improve self-confidence by guiding elderly diabetic patients to reflect on past self-management challenges and share successful self-management experiences. At the same time, learn how to find self-management problems, set goals and develop action plans, and other strategies to help elderly patients with diabetes set goals for their own health problems, develop and implement self-suitable, feasible and sustainable self-management behaviors to strengthen Self-management skills for elderly diabetic patients. The 4-week program was implemented for 2 hours/week.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years,older adult peer leaders with diabetes, elementary school or higher level of education,

Exclusion Criteria:

* People with cognitive impairment, severe diabetes complications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1C | Change from Baseline HbA1C at 3 months
  Hemoglobin A1c, HbA1c

SECONDARY OUTCOMES:
Self-Management Score | Change from Baseline Self-Management Score at 3 months
  Diabetes Self-Management Instrument Short Form, DSMI-20
Self-Efficacy Score | Change from Baseline Self-Efficacy Score at 3 months
  The Diabetes Management Self-Efficacy Scale, DMSES

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chun Chen, Master, Study Chair — St. Martin De Porres Hospital
Locations (1):
- St. Martin De Porres Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD for study protocol
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: Email Request

REFERENCES:
- [Derived] Chen WC, Kuo CC, Lin CC, Wu CC. A preliminary study on the effects of the Peer-Led Self-Management (PLSM) program on self-efficacy, self-management, and physiological measures in older adults with diabetes: A block randomized controlled trial. Geriatr Nurs. 2021 Mar-Apr;42(2):386-396. doi: 10.1016/j.gerinurse.2021.01.011. Epub 2021 Feb 20. PMID 33621782
- [Derived] Chen WC, Lin CC, Kuo CC, Wu CC, Liu TJ, Chen MT. A Theory-Based Self-Management Training Program for Older Adult Peer Leaders with Diabetes: A Feasibility Assessment. J Multidiscip Healthc. 2021 Jan 7;14:33-44. doi: 10.2147/JMDH.S286186. eCollection 2021. PMID 33442261